CLINICAL TRIAL: NCT01257828
Title: Efficacy of Riluzole in Patients With Cervical Spondylotic Myelopathy Undergoing Surgical Treatment. A Randomized, Double-Blind, Placebo-controlled Multi-Center Study
Brief Title: Efficacy of Riluzole in Surgical Treatment for Cervical Spondylotic Myelopathy (CSM-Protect)
Acronym: CSM-Protect
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOSpine North America Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPN-10-001
Record Dates: First submitted 2010-10-23; First posted 2010-12-10 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Cervical Spondylotic Myelopathy
MeSH Terms: interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo medication and decompressive cervical spine surgery
  Interventions: Drug: Placebo medication
- Riluzole (Experimental): Riluzole in dose 50mg BID for 14 days prior to surgery and 28 days after the decompressive spine surgery
  Interventions: Drug: riluzole

INTERVENTIONS:
Drug: riluzole — 50mg BID orally for 14 days prior to surgery and 28 days after the surgery
  Other Names: Rilutek
  Arms: Riluzole
Drug: Placebo medication — 50mg BID orally for 14 days prior to surgery and 28 days after the surgery
  Arms: Placebo

SUMMARY:
CSM (Cervical spondylotic myelopathy) is the most common cause of spinal cord injury worldwide. While there is evidence from the recently completed SpineNet prospective study that surgical decompression is an effective treatment for CSM, it is clear that many patients have remaining neurological impairment. While surgery is relatively safe, approximately 3% of patients maintain a neurological problem. Given this background and data from preclinical models of non-traumatic and traumatic spinal cord injury, there is strong evidence to consider the potential benefit of adding a neuroprotective drug which aids in the treatment of patients with CSM whom are undergoing surgical decompression. Riluzole is FDA-approved for the treatment of amyotrophic lateral sclerosis, which has some similar clinical features to CSM. Riluzole is currently under investigation for traumatic spinal cord injury. Given this background, there is a strong basis to consider studying the potential neurological benefits of Riluzole as a treatment to surgical decompression in patients with CSM.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Diagnosis of symptomatic cervical spondylotic myelopathy defined as a combination of:

  1. one or more of the following symptoms:

     * Numb hands
     * Clumsy hands
     * Impairment of gait
     * Bilateral arm paresthesiae
     * l'Hermitte's phenomena
     * Weakness And,
  2. one or more of the following signs:

     * Corticospinal distribution motor deficits
     * Atrophy of hand intrinsic muscles
     * Hyperreflexia
     * Positive Hoffman sign
     * Upgoing plantar responses
     * Lower limb spasticity
     * Broad based, unstable gait And,
  3. MRI evidence of cervical spondylotic myelopathy
* Scheduled for an elective surgery for cervical spondylotic myelopathy
* Preoperative mJOA score ≥8 and ≤14
* Women of child bearing potential must be:

  * Postmenopausal defined as amenorrhea for at least 2 years.
  * Surgically sterile, (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy)
  * Abstinent (at the discretion of the investigator)
  * Having other congenital or medical condition that prevents subject from becoming pregnant
  * If sexually active, be practicing an effective method of birth control such as hormonal prescription oral contraceptives, progesterone implants or injections, intrauterine device (IUD), or male partner with a vasectomy. A double-barrier method such as condoms, diaphragms or cervical caps with spermicidal foam, cream or gel may be used as a birth control method.
  * Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test or a negative urine pregnancy test at screening before the first dose of study drug is received.

Exclusion Criteria:

* Previous surgery for CSM
* Concomitant symptomatic lumbar stenosis
* CSM symptoms due to cervical trauma (at the discretion of the investigator)
* Hypersensitivity to riluzole or any of its components
* Neutropenia measured as absolute neutrophil count (ANC) measured in cells per microliter of blood of < 1500 at screening visit
* Creatinine level of > 1.2 milligrams (mg) per deciliter (dl) in males or > 1.1 milligrams per deciliter in females at screening visit Liver enzymes (ALT or AST) 3x higher than normal values at screening visit.
* Liver enzymes (ALT or AST) 3x higher than normal values at screening visit.
* Subject will be using any of the following medications which are classified as CYP1A2 inhibitors or inducers*during the course of the drug regimen:

Inhibitors:

* Ciprofloxacin
* Enoxacin
* Fluvoxamine
* Methoxsalen
* Mexiletine
* Oral contraceptives
* Phenylpropanolamine
* Thiabendazole
* Zileuton

Inducers:

* Montelukast
* Phenytoin

  *Note: no washout period required; if these medications are discontinued, subjects are eligible to be enrolled in the trial.
* Systemic infection such as AIDS, HIV, and active hepatitis
* Active malignancy defined as history of invasive malignancy, except if the patient has received treatment and displayed no clinical signs and symptoms for at least five years
* Recent history (less than 3 years) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation
* Breastfeeding at screening visit and plan to continue during the course of the study drug
* Unlikely to comply with the follow-up evaluation schedule
* Unlikely to comply with investigational drug regime
* Participation in a clinical trial of another investigational drug or device within the past 30 days
* Is a prisoner
* Unable to converse, read or write English at elementary school level

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Modified Japanese Orthopedic Association Score (mJOA) | Before the surgery, 180 days
  The mJOA is a clinician administered scale. It evaluates four clinical dimensions; motor dysfunction score for upper and lower extremities, sensation loss and sphincter dysfunction. The total score ranges from 0 (worst) to 18 (best).

SECONDARY OUTCOMES:
Nurick Score | Pre-surgical, 180 days
  Nurick score is a simple measure of neurological dysfunction and ranges from 0 (best) to 6 (worst).
SF-36v2.0 | Before the surgery, 180 days
  The SF36v2.0 is a health-related quality of life instrument that evaluates health status accross eight health dimensions.
Neck Disability Index (NDI) | Before the surgery, 180 days
  The NDI evaluates patient self-reported functional outcomes related to neck conditions. The NDI score ranges from 0 (best) to 100 (worst).
Cervical Pain Numeric Rating Scale | Before the surgery, 180 days
  Simple numeric rating scale with choises of answers from 0 (no pain) to 10 (worst imaginable pain)
EQ-5D | Before the surgery, 180 days
  EQ-5D™ is a standardised instrument for use as a measure of health outcome. It provides a simple descriptive profile and a single index value for health status.
American Spinal Injury Association Score (ASIA) | Before the surgery, 180 days
  The ASIA impairment scale describes a person's functional impairment as a result of their spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fehlings, MD, Principal Investigator — University Health Network, Toronto; Branko Kopjar, MD, Study Director — University of Washington
Locations (21):
- United States (15):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC Davis Spine Center, Sacramento, California
  - University of California - San Francisco, San Francisco, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Louisiana State University, Baton Rouge, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Orthopaedics, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Rothman Institute Orthopaedics, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - St. Michael's Hospital, Toronto, Ontario
  - University of Toronto Hospital, Toronto, Ontario
  - McGill University Health Centre, Montral, Quebec
  - Montreal Neurological Institute, Montreal, Quebec
  - University of Saskatchewan, Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Fehlings MG, Wilson JR, Karadimas SK, Arnold PM, Kopjar B. Clinical evaluation of a neuroprotective drug in patients with cervical spondylotic myelopathy undergoing surgical treatment: design and rationale for the CSM-Protect trial. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S68-75. doi: 10.1097/BRS.0b013e3182a7e9b0. PMID 23962993
- [Derived] Bak AB, Moghaddamjou A, Arnold PM, Harrop JS, Fehlings MG. Chronic pain after decompression for degenerative cervical myelopathy: a pooled trajectory analysis of individual participant data. Pain. 2025 Oct 15. doi: 10.1097/j.pain.0000000000003828. Online ahead of print. PMID 41086299
- [Derived] Wong R, Alvi MA, Quddusi AI, Fehlings MG. Role of Neck Pain in Defining Clinical Trajectories of Outcomes in Patients With Degenerative Cervical Myelopathy: Results of a Novel Machine Learning Algorithm. Global Spine J. 2025 May 10;16(1):21925682251341263. doi: 10.1177/21925682251341263. Online ahead of print. PMID 40347099
- [Derived] Pedro KM, Alvi MA, Hejrati N, Moghaddamjou A, Fehlings MG. Elderly Patients Show Substantial Improvement in Health-Related Quality of Life After Surgery for Degenerative Cervical Myelopathy Despite Medical Frailty: An Ambispective Analysis of a Multicenter, International Data Set. Neurosurgery. 2024 Jan 10. doi: 10.1227/neu.0000000000002818. Online ahead of print. PMID 38197642
- [Derived] Fehlings MG, Badhiwala JH, Ahn H, Farhadi HF, Shaffrey CI, Nassr A, Mummaneni P, Arnold PM, Jacobs WB, Riew KD, Kelly M, Brodke DS, Vaccaro AR, Hilibrand AS, Wilson J, Harrop JS, Yoon ST, Kim KD, Fourney DR, Santaguida C, Massicotte EM, Kopjar B. Safety and efficacy of riluzole in patients undergoing decompressive surgery for degenerative cervical myelopathy (CSM-Protect): a multicentre, double-blind, placebo-controlled, randomised, phase 3 trial. Lancet Neurol. 2021 Feb;20(2):98-106. doi: 10.1016/S1474-4422(20)30407-5. Epub 2020 Dec 22. PMID 33357512